CLINICAL TRIAL: NCT04307641
Title: Strengthening Patient-Centered Accessibility, Respect, and Quality of Care for Abortion Clients in UP, India
Brief Title: Improving Person Centered Care for Abortion Clients in India
Acronym: SPARQ_ACI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Public Health Foundation of India (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 15-18008_India Abortion
Record Dates: First submitted 2020-03-10; First posted 2020-03-13 (Actual); Last update posted 2023-05-24 (Actual); Status verified 2020-03

CONDITIONS: Reproductive Health
Keywords: abortion; person-centered care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Pharmacists who received in the intervention.
  Interventions: Behavioral: 2 Page Information Sheet
- Control (No Intervention): Pharmacists who did not received in the intervention.

INTERVENTIONS:
Behavioral: 2 Page Information Sheet — 2 page information sheet about medication abortion
  Arms: Intervention

SUMMARY:
The purpose of this study is to understand the effect of providing pharmacists in UP, India with additional information about medication abortion.

DETAILED DESCRIPTION:
This study evaluates whether providing pharmacists with additional information about medication abortion can improve abortion person-centered care for women accessing MA at these sites.

ELIGIBILITY:
Inclusion Criteria:

* Pharmacist providing medication abortion within Lucknow, Kanpur, Unnao
* Agreed to participate

Exclusion Criteria:

* Pharmacists not providing medication abortion within Lucknow, Kanpur, Unnao
* Did not agree to participate

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 283 (Actual)
Dates: Start 2016-11-01 (Actual); Primary Completion 2018-07-01 (Actual); Study Completion 2018-07-01 (Actual)

PRIMARY OUTCOMES:
Change in knowledge about medication abortion | baseline compared to 6-months after intervention
  self-reported survey (dose, time, side effects, complications)

SECONDARY OUTCOMES:
Provider behavior when providing medication abortion (MA) to clients | 3-months post intervention
  Information provided to mystery clients regarding MA (dose, time, side effects, complications)
Interest and satisfaction with intervention | 6-months after intervention
  self-reported survey on interest and satisfaction

CONTACTS AND LOCATIONS:
Overall Officials: Nadia Diamond-Smith, PhD, Principal Investigator — University of California, San Francisco

IPD SHARING:
Plan to Share IPD: Yes
The data from this evaluation will be shared on the data repository Dryad.
Time Frame: Data will be made available following the publication of the first journal article based on this data.
Access Criteria: Anyone who has access to Dryad